CLINICAL TRIAL: NCT05266456
Title: A Phase 1/2, Randomized, Observer-Blind, Dose-Finding, Controlled, Parallel-Group, Two-Stage Clinical Study to Evaluate the Safety, Tolerability, and Immunogenicity of a 24-Valent Pneumococcal Conjugate Vaccine (VAX-24) in Healthy Adults Aged 18 to 64 Years
Brief Title: Safety, Tolerability, and Immunogenicity Study of a 24-Valent Pneumococcal Conjugate Vaccine (VAX-24) in Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vaxcyte, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAX24-101
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-03

CONDITIONS: Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- VAX-24 Low Dose (Experimental): Participants will receive a single dose of VAX-24 1.1 mcg administered as an intramuscular injection on Day 1.
  Interventions: Biological: 24 valent pneumococcal conjugate vaccine
- VAX-24 Mid Dose (Experimental): Participants will receive a single dose of VAX-24 2.2 mcg administered as an intramuscular injection on Day 1.
  Interventions: Biological: 24 valent pneumococcal conjugate vaccine
- VAX-24 Mixed Dose (Experimental): Participants will receive a single dose of VAX-24 2.2 mcg/4.4 mcg administered as an intramuscular injection on Day 1.
  Interventions: Biological: 24 valent pneumococcal conjugate vaccine
- PCV20 (Active Comparator): Participants will receive a single intramuscular injection of the standard dose of PCV20 on Day 1.
  Interventions: Biological: 20 valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 24 valent pneumococcal conjugate vaccine — 0.5 ml dose of VAX-24 will be administered into the deltoid muscle at Day 1
  Arms: VAX-24 Low Dose; VAX-24 Mid Dose; VAX-24 Mixed Dose
Biological: 20 valent pneumococcal conjugate vaccine — 0.5 ml dose of PCV20 will be administered into the deltoid muscle at Day 1
  Arms: PCV20

SUMMARY:
The objective of the study is to evaluate the safety and tolerability of a single injection of VAX-24 at 3 dose levels compared to Prevnar 20™ (PCV20) in adults 18 to 49 years of age in Phase 1. The Phase 2 will evaluate the safety, tolerability, and immunogenicity of a single injection of VAX-24 at 3 dose levels compared to PCV20 in adults aged 50 to 64 years of age in Phase 2.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the safety and tolerability of a single injection of VAX-24 at 3 dose levels (Low: 1.1 mcg; Mid: 2.2 mcg; or Mixed: 2.2/4.4 mcg) compared to Prevnar 20™ (PCV20) in adults 18 to 49 years of age in Phase 1. The Phase 2 will evaluate the safety, tolerability, and immunogenicity of a single injection of VAX-24 at 3 dose levels (Low: 1.1 mcg; Mid: 2.2 mcg; or Mixed: 2.2/4.4 mcg) compared to PCV20 in adults aged 50 to 64 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 to 49 years (inclusive) for the Phase 1 group, or 50 to 64 years (inclusive) for the Phase 2 group at the time of enrollment into the study.
* Able and willing to complete the informed consent process.
* Available for clinical follow-up through the last study visit at 6 months after the study vaccination.
* In good general health as determined by medical history, vital signs, physical examination, and clinical judgment of the investigator.
* Screening laboratory values must be within the central laboratory normal limits prior to study enrollment. Minor abnormalities are considered acceptable if not clinically significant.
* Willing to have blood samples collected, stored indefinitely, and used for research purposes.
* Able to provide proof of identity to the satisfaction of the study staff completing the enrollment process.
* Negative pregnancy test (urine and serum) for women of childbearing potential.

Exclusion Criteria:

* Previous pneumococcal disease (either confirmed or by self-reporting).
* Previous receipt of a licensed or investigational pneumococcal vaccine.
* Receipt of any investigational study product within 30 days prior to enrollment into the study, currently participating in another interventional investigational study, or having plans to receive another investigational product(s) while on study.
* Planned or actual administration of any licensed vaccine during the period starting 30 days before enrollment into the study through Day 29.
* Physical examination indicating any clinically significant medical condition.
* Body Temperature > 38.0°C (> 100.4°F) or acute illness within 3 days prior to study vaccination (subject may be rescheduled).
* Seropositive to HIV, HCV, or HBsAg.
* History of severe allergic reaction with generalized urticaria, angioedema, or anaphylaxis.
* Female who is breast-feeding or planning to become pregnant during study participation.
* Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
* Any other chronic or clinically significant medical condition that, in the opinion of the investigator, would jeopardize the safety or rights of the subject or confound evaluation of the study vaccine.
* Any medical, psychiatric, or social condition that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a subject's ability to give informed consent.
* Received blood or blood product (including Immune Globulin IV) within 90 days prior to enrollment into the study.
* Received systemic corticosteroids for ≥ 14 consecutive days and has not completed treatment ≤30 days prior to enrollment into the study.
* Receiving immunosuppressive therapy.
* History of malignancy ≤5 years before enrollment, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 835 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Vaxcyte, Inc.
Locations (13):
- United States (13):
  - CenExel RCA, Hollywood, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Meridian Clinical Research, Savannah, Georgia
  - Velocity Clinical Research, Valparaiso, Indiana
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Benchmark Research, Metairie, Louisiana
  - Alliance for Multispecialty Research, Kansas City, Missouri
  - Rochester Clinical Research, Rochester, New York
  - Acellacare of Wilmington, Wilmington, North Carolina
  - Velocity Clinical Research, Warwick, Rhode Island
  - Coastal Carolina Research, North Charleston, South Carolina
  - Benchmark Research, San Angelo, Texas
  - JBR Clinical Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Vaxcyte is committed to providing access to anonymized data from the company's clinical trials for the purpose of legitimate scientific research. Requests for data may be addressed to datasharing@vaxcyte.com. Requests must be accompanied by a detailed analysis plan and will be reviewed for scientific validity. Data will be made available after initial product approval. Sharing of data may require execution of a data-sharing agreement.
Supporting Information: Study Protocol
Time Frame: Individual participant data will be shared after deidentification and made available starting 6 months after initial product approval.
Access Criteria: Criteria will depend on the specific proposal received and may include qualification of the scientific researchers, potential contribution to the research field, scientific rigor of statistical and analytical methods, and other criteria appropriate for the proposal.

REFERENCES:
- [Result] Wassil J, Sisti M, Fairman J, Davis M, Fierro C, Bennett S, Johnson D, Migone TS, Nguyen K, Sauer P, Currie M, Iki S, Simon JK. Evaluating the safety, tolerability, and immunogenicity of a 24-valent pneumococcal conjugate vaccine (VAX-24) in healthy adults aged 18 to 64 years: a phase 1/2, double-masked, dose-finding, active-controlled, randomised clinical trial. Lancet Infect Dis. 2024 Mar;24(3):308-318. doi: 10.1016/S1473-3099(23)00572-8. Epub 2023 Dec 4. PMID 38061367

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject was enrolled 22-Feb-2022 and last subject randomized/vaccinated was 01-Jul-22. Study sites were medical clinics.
Pre-assignment Details: In Phase 1, 95 participants were screened; 21 did not meet inclusion/exclusion criteria, 4 withdrew consent, and 6 discontinued for other reason. Five of Phase 1 screen failures were rescreened and enrolled in Phase 2. An additional 1001 participants were screened (for a total of 1006); of these, 235 failed screening: 173 did not meet inclusion/exclusion criteria, 12 withdrew consent, and 50 failed for other reasons.
Groups:
- VAX-24 Low Dose: Participants will receive a single dose of VAX-24 administered as an intramuscular injection on Day 1 at the 1.1 mcg dose levels.
  24 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-24 will be administered into the deltoid muscle at Day 1
- VAX-24 Mid Dose: Participants will receive a single dose of VAX-24 administered as an intramuscular injection on Day 1 at 2.2 mcg dose level.
  24 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-24 will be administered into the deltoid muscle at Day 1
- VAX-24 Mixed Dose: Participants will receive a single dose of VAX-24 administered as an intramuscular injection on Day 1 at 2.2/4.4 mcg dose levels.
  24 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-24 will be administered into the deltoid muscle at Day 1
Period: Phase 1, Adults 18-49 Years of Age
Arm/Group | VAX-24 Low Dose | VAX-24 Mid Dose | VAX-24 Mixed Dose | PCV20
Started | 16 | 16 | 16 | 16
Completed | 15 | 15 | 16 | 15
Not Completed | 1 | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Period: Phase 2, Adults 50-64 Years
Arm/Group | VAX-24 Low Dose | VAX-24 Mid Dose | VAX-24 Mixed Dose | PCV20
Started | 193 | 192 | 192 | 194
Completed | 186 | 186 | 187 | 192
Not Completed | 7 | 6 | 5 | 2
Not completed — Lost to Follow-up | 6 | 6 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0
Not completed — Unavailable for follow up | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline demographics include all randomized subjects from Phase 1 and Phase 2 by age group. The prespecified immunogenicity analysis and Laboratory Value Abnormalities and/or Potentially Clinically Significant Laboratory Values included only subjects 50-64 years old.
Groups:
- VAX-24 Low Dose 18-49 Yrs; VAX-24 Low Dose 50-64 Yrs: Participants will receive a single dose of VAX-24 administered as an intramuscular injection on Day 1 at 1.1 mcg dose level.
  24 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-24 will be administered into the deltoid muscle at Day 1
- VAX-24 Mid Dose 18-49 Yrs; VAX-24 Mid Dose 50-64 Yrs: Participants will receive a single dose of VAX-24 administered as an intramuscular injection on Day 1 at 2.2 mcg dose level.
  24 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-24 will be administered into the deltoid muscle at Day 1
- VAX-24 Mixed Dose 18-49 Yrs; VAX-24 Mixed Dose 50-64 Yrs: Participants will receive a single dose of VAX-24 administered as an intramuscular injection on Day 1 at 2.2 mcg/4.4 mcg dose levels.
  24 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-24 will be administered into the deltoid muscle at Day 1
- PCV20 18-49 Yrs; PCV20 50-64 Yrs: Participants will receive a single intramuscular injection of the standard dose of PCV20 on Day 1.
  20 valent pneumococcal conjugate vaccine: 0.5 ml dose of PCV20 will be administered into the deltoid muscle at Day 1
- Total: Total of all reporting groups
Arm/Group | VAX-24 Low Dose 18-49 Yrs | VAX-24 Mid Dose 18-49 Yrs | VAX-24 Mixed Dose 18-49 Yrs | PCV20 18-49 Yrs | VAX-24 Low Dose 50-64 Yrs | VAX-24 Mid Dose 50-64 Yrs | VAX-24 Mixed Dose 50-64 Yrs | PCV20 50-64 Yrs | Total
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 193 | 192 | 192 | 194 | 835
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 39.5 [35.0 to 46.5] | 34.0 [30.0 to 37.5] | 39.0 [28.5 to 43.0] | 37.0 [26.5 to 41.5] | 57.0 [53.0 to 60.0] | 57.0 [53.5 to 60.0] | 57.0 [53.0 to 60.0] | 57.0 [53.0 to 60.0] | 57.0 [53.0 to 60.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 8 | 8 | 110 | 121 | 134 | 127 | 522
  Male | 9 | 9 | 8 | 8 | 83 | 71 | 58 | 67 | 313
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 2 | 3 | 22 | 18 | 22 | 17 | 93
  Not Hispanic or Latino | 12 | 10 | 14 | 13 | 171 | 172 | 168 | 177 | 737
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3
  Asian | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 5 | 7 | 4 | 10 | 40 | 32 | 29 | 29 | 156
  White | 10 | 8 | 12 | 4 | 145 | 157 | 156 | 154 | 646
  More than one race | 1 | 0 | 0 | 0 | 2 | 1 | 4 | 3 | 11
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 3 | 2 | 1 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 16 | 16 | 193 | 192 | 192 | 194 | 835
Height (cm) [Median (Inter-Quartile Range); unit: cm] | 176.1 [166.3 to 183.3] | 170.1 [165.1 to 179.2] | 167.1 [161.2 to 188.0] | 170.8 [165.1 to 176.6] | 168.3 [162.6 to 176.5] | 167.6 [162.6 to 175.3] | 167.6 [160.6 to 173.0] | 167.6 [160.0 to 176.5] | 167.6 [161.3 to 175.8]
Weight (kg) [Median (Inter-Quartile Range); unit: kg] | 80.85 [69.91 to 96.16] | 92.10 [74.94 to 117.24] | 90.50 [71.96 to 103.65] | 78.07 [72.04 to 96.62] | 87.82 [71.85 to 103.42] | 86.72 [72.58 to 104.33] | 83.10 [70.46 to 97.39] | 82.83 [70.31 to 97.52] | 84.81 [71.67 to 99.97]
Body Mass Index (kg/m^2) Median, Q1 - Q3 [Median (Inter-Quartile Range); unit: kg/m^2] | 26.99 [24.01 to 30.12] | 31.09 [26.20 to 36.81] | 29.16 [26.66 to 34.56] | 26.91 [23.95 to 31.83] | 29.87 [25.75 to 35.99] | 30.65 [26.15 to 35.88] | 29.34 [25.20 to 33.20] | 29.06 [25.41 to 34.28] | 29.49 [25.61 to 34.68]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Solicited Local Reactions Within 7 Days After Vaccination in Each Age Group
Description: Solicited local reactions include redness/erythema, swelling/induration, and pain at injection site within 7 days after vaccination in each age group
Time Frame: 7 days after vaccination
Population: Safety population, defined as all patients exposed to study vaccine. Subject safety data were analyzed according to the vaccine regimen they received: 1 subject was randomized to VAX-24 2.2/4.4 mcg but received VAX-24 2.2 mcg, and 2 subjects were randomized to VAX-24 2.2 mcg but received PCV20.
Measure: Number; unit: percentage of participants
Groups:
- VAX-24 Low Dose 18-49 Yrs; VAX-24 Low Dose 50-64 Yrs; VAX24 Low Dose 18-64 Yrs: Participants will receive a single dose of VAX-24 administered as an intramuscular injection on Day 1 at 1.1 mcg dose levels.
  24 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-24 will be administered into the deltoid muscle at Day 1
- VAX-24 Mid Dose 18-64 Yrs: Participants will receive a single dose of VAX-24 administered as an intramuscular injection on Day 1 at 2.2 mcg dose levels.
  24 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-24 will be administered into the deltoid muscle at Day 1
- VAX-24 Mixed Dose 18-64 Yrs: Participants will receive a single dose of VAX-24 administered as an intramuscular injection on Day 1 at 2.2 mcg/4.4 mcg dose levels.
  24 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-24 will be administered into the deltoid muscle at Day 1
- PCV20 18-64 Yrs: Participants will receive a single intramuscular injection of the standard dose of PCV20 on Day 1.
  20 valent pneumococcal conjugate vaccine: 0.5 ml dose of PCV20 will be administered into the deltoid muscle at Day 1
Arm/Group | VAX-24 Low Dose 18-49 Yrs | VAX-24 Mid Dose 18-49 Yrs | VAX-24 Mixed Dose 18-49 Yrs | PCV20 18-49 Yrs | VAX-24 Low Dose 50-64 Yrs | VAX-24 Mid Dose 50-64 Yrs | VAX-24 Mixed Dose 50-64 Yrs | PCV20 50-64 Yrs | VAX24 Low Dose 18-64 Yrs | VAX-24 Mid Dose 18-64 Yrs | VAX-24 Mixed Dose 18-64 Yrs | PCV20 18-64 Yrs
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 193 | 191 | 191 | 196 | 209 | 207 | 207 | 212
percentage of participants
  Any solicited local AE; Overall, Any Grade | 56.3 | 81.3 | 81.3 | 93.8 | 73.6 | 71.7 | 77.5 | 71.9 | 72.2 | 72.5 | 77.8 | 73.6
  Pain at injection site; Overall, Any Grade | 56.3 | 75.0 | 81.3 | 81.3 | 71.0 | 71.2 | 77.0 | 69.9 | 69.9 | 71.5 | 77.3 | 70.8
  Erythema (redness) at injection site; Overall, Any Grade | 6.3 | 6.3 | 18.8 | 25.0 | 6.7 | 7.9 | 8.9 | 8.7 | 6.7 | 7.7 | 9.7 | 9.9
  Edema (swelling) at injection site; Overall, Any Grade | 18.8 | 12.5 | 25.0 | 18.8 | 8.8 | 7.9 | 7.9 | 10.7 | 9.6 | 8.2 | 9.2 | 11.3

2. Primary Outcome: Percentage of Participants Reporting Solicited Systemic Events Within 7 Days After Vaccination in Each Age Group
Description: Solicited systemic reactions include fever, headache, fatigue, muscle pain, and joint pain
Time Frame: 7 days after vaccination
Population: Safety population, which included all subjects in the Exposed Population who provided safety assessment data. Subject safety data were analyzed according to the vaccine regimen they received: 1 subject was randomized to VAX-24 2.2/4.4 mcg but received VAX-24 2.2 mcg, and 2 subjects were randomized to VAX-24 2.2 mcg but received PCV20.
Measure: Number; unit: Percentage of participants
Groups:
- VAX-24 Low Dose 18-64 Yrs: Participants will receive a single dose of VAX-24 administered as an intramuscular injection on Day 1 at 1.1 mcg dose level.
  24 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-24 will be administered into the deltoid muscle at Day 1
- VAX-24 Mid Dose 18-64 Yrs: Participants will receive a single dose of VAX-24 administered as an intramuscular injection on Day 1 at 2.2 mcg dose level.
  24 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-24 will be administered into the deltoid muscle at Day 1
Arm/Group | VAX-24 Low Dose 18-49 Yrs | VAX-24 Mid Dose 18-49 Yrs | VAX-24 Mixed Dose 18-49 Yrs | PCV20 18-49 Yrs | VAX-24 Low Dose 50-64 Yrs | VAX-24 Mid Dose 50-64 Yrs | VAX-24 Mixed Dose 50-64 Yrs | PCV20 50-64 Yrs | VAX-24 Low Dose 18-64 Yrs | VAX-24 Mid Dose 18-64 Yrs | VAX-24 Mixed Dose 18-64 Yrs | PCV20 18-64 Yrs
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 193 | 191 | 191 | 196 | 209 | 207 | 207 | 212
Percentage of participants
  Any solicited systemic adverse event | 50.0 | 62.5 | 56.3 | 75.0 | 69.4 | 69.6 | 71.2 | 64.8 | 67.9 | 69.1 | 70.0 | 65.6
  Fever (oral temperature >= 100.4ºF) | 6.3 | 6.3 | 0.0 | 12.5 | 1.0 | 0.5 | 2.1 | 1.0 | 1.4 | 1.0 | 1.9 | 1.9
  Fatigue | 37.5 | 31.3 | 37.5 | 50.0 | 42.5 | 40.8 | 40.8 | 39.8 | 42.1 | 40.1 | 40.6 | 40.6
  Headache | 31.3 | 37.5 | 25.0 | 37.5 | 30.6 | 28.8 | 30.4 | 30.1 | 30.6 | 29.5 | 30.0 | 30.7
  Muscle Pain | 37.5 | 37.5 | 18.8 | 56.3 | 57.0 | 56.0 | 60.2 | 53.1 | 55.5 | 54.6 | 57.0 | 53.3
  Joint Pain | 25.0 | 12.5 | 12.5 | 43.8 | 24.9 | 16.2 | 27.7 | 24.0 | 24.9 | 15.9 | 26.6 | 25.5

3. Primary Outcome: Percentage of Participants Reporting Unsolicited Adverse Events (AE) in Each Age Group
Description: Percentage of participants in each age group with adverse events (AEs) whose date of onset occurs after the study vaccine and within the 28 days after vaccination.
Time Frame: 1 month after vaccination
Population: Safety population, including all subjects in the Exposed Population who provided safety assessment data. Subject safety data were analyzed according to the vaccine regimen they received: 1 subject was randomized to VAX-24 2.2/4.4 mcg but received VAX-24 2.2 mcg, and 2 subjects were randomized to VAX-24 2.2 mcg but received PCV20.
Measure: Number; unit: Percentage of participants
Groups:
- VAX-24 Mixed Dose 18-49 Yrs; VAX-24 Mixed Dose 18-64 Yrs: Participants will receive a single dose of VAX-24 administered as an intramuscular injection on Day 1 at 2.2/4.4 mcg dose levels.
  24 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-24 will be administered into the deltoid muscle at Day 1
- VAX-24 Mid Dose 50-64 Yrs: Participants will receive a single dose of VAX-24 administered as an intramuscular injection on Day 1 at 2.2 mcg dose levels.
  24 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-24 will be administered into the deltoid muscle at Day 1
- PCV20 50-64; PCV20 18-64 Yrs: Participants will receive a single intramuscular injection of the standard dose of PCV20 on Day 1.
  20 valent pneumococcal conjugate vaccine: 0.5 ml dose of PCV20 will be administered into the deltoid muscle at Day 1
- VAX-24 Low Dose 18-64: Participants will receive a single dose of VAX-24 administered as an intramuscular injection on Day 1 at 1.1 mcg dose levels.
  24 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-24 will be administered into the deltoid muscle at Day 1
Arm/Group | VAX-24 Low Dose 18-49 Yrs | VAX-24 Mid Dose 18-49 Yrs | VAX-24 Mixed Dose 18-49 Yrs | PCV20 18-49 Yrs | VAX-24 Low Dose 50-64 Yrs | VAX-24 Mid Dose 50-64 Yrs | VAX-24 Mixed Dose 50-64 Yrs | PCV20 50-64 | VAX-24 Low Dose 18-64 | VAX-24 Mid Dose 18-64 Yrs | VAX-24 Mixed Dose 18-64 Yrs | PCV20 18-64 Yrs
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 193 | 191 | 191 | 196 | 209 | 207 | 207 | 212
Percentage of participants | 12.5 | 12.5 | 6.3 | 6.3 | 15.5 | 11.5 | 13.1 | 16.8 | 15.3 | 11.6 | 12.6 | 16.0

4. Primary Outcome: Percentage of Participants Reporting SAEs and New Onset of Chronic Illnesses (NOCI)
Description: Percentage of participants with SAEs and NOCIs
Time Frame: 6 months after vaccination
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Groups:
- VAX-24 Mixed Dose; VAX-24 Mixed Dose 18-64 Yrs: Participants will receive a single dose of VAX-24 administered as an intramuscular injection on Day 1 at 2.2 mcg/4.4 mcg dose levels.
  24 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-24 will be administered into the deltoid muscle at Day 1
Arm/Group | VAX-24 Low Dose 18-49 Yrs | VAX-24 Mid Dose 18-49 Yrs | VAX-24 Mixed Dose 18-49 Yrs | PCV20 18-49 Yrs | VAX-24 Low Dose 50-64 Yrs | VAX-24 Mid Dose 50-64 Yrs | VAX-24 Mixed Dose | PCV20 50-64 Yrs | VAX-24 Low Dose 18-64 Yrs | VAX-24 Mid Dose 18-64 Yrs | VAX-24 Mixed Dose 18-64 Yrs | PCV20 18-64 Yrs
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 193 | 191 | 191 | 196 | 209 | 207 | 207 | 212
percentage of participants
  Subjects with at least one SAE | 0 | 0 | 0 | 0 | 1.0 | 1.6 | 0.5 | 2.0 | 1.0 | 1.4 | 0.5 | 1.9
  Subjects with at least one NOCI | 0 | 0 | 0 | 0 | 1.6 | 1.6 | 3.1 | 2.6 | 1.4 | 1.4 | 2.9 | 2.4

5. Secondary Outcome: Percentage of Participants With Laboratory Value Abnormalities and/or Potentially Clinically Significant Laboratory Values
Description: Shifts from Normal at Baseline to Abnormal on Day 29 in Clinical Chemistry Parameters Occurring in >5% of Subjects Aged 50 to 64 Years
Time Frame: 1 month after vaccination
Population: Prespecified analysis population included all subjects age 50-64 in the Exposed Population who provided safety assessment data. Subject safety data were analyzed according to the vaccine regimen they received: 1 subject was randomized to VAX-24 2.2/4.4 mcg but received VAX-24 2.2 mcg, and 2 subjects were randomized to VAX-24 2.2 mcg but received PCV20.
Measure: Number; unit: percentage of participants
Groups:
- VAX-24 Low Dose: Participants will receive a single dose of VAX-24 administered as an intramuscular injection on Day 1 at 1.1 mcg dose level.
  24 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-24 will be administered into the deltoid muscle at Day 1
Arm/Group | VAX-24 Low Dose | VAX-24 Mid Dose | VAX-24 Mixed Dose | PCV20
Number analyzed (Participants) | 193 | 191 | 191 | 196
percentage of participants
  Bicarbonate: Low | 14.4 | 18.4 | 15.0 | 11.8
  Cholesterol: High | 7.2 | 7.7 | 8.7 | 8.5
  Triglycerides: High | 9.1 | 8.2 | 9.7 | 10.8
  Creatinine: High | 11.5 | 11.1 | 10.6 | 8.5
  Glucose: High | 7.2 | 3.9 | 5.3 | 7.1
  Uric Acid: High | 8.1 | 7.2 | 2.9 | 5.7

6. Secondary Outcome: VAX-24 Pneumococcal Serotype-specific Opsonophagocytic Assay (OPA) Geometric Mean Titer (GMTs)
Description: Antibody geometric mean titers as measured by OPA for the 24 pneumococcal serotypes in VAX-24
Time Frame: 1 month after vaccination
Population: Prespecified Immunogenicity Evaluable Population included all subjects 50 to 64 years in the Exposed Population with no major protocol deviation impacting immunogenicity assessment, no prohibited medication or vaccine, and provided evaluable serum sample results for baseline and Day 29 within required time frames. Data were analyzed according to vaccine received: 1 subject randomized to VAX-24 2.2/4.4 mcg received VAX-24 2.2 mcg; 2 subjects randomized to VAX-24 2.2 mcg received PCV20.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | VAX-24 Low Dose | VAX-24 Mid Dose | VAX-24 Mixed Dose | PCV20
Number analyzed (Participants) | 193 | 191 | 191 | 196
Titer
  1: number analyzed (Participants) | 164 | 176 | 169 | 177
  1 | 190.08 [147.05 to 245.69] | 317.62 [246.32 to 409.56] | 228.09 [176.35 to 295.01] | 358.18 [278.29 to 461.00]
  2: number analyzed (Participants) | 163 | 177 | 170 | 177
  2 | 1371.45 [1135.70 to 1656.12] | 1698.18 [1409.82 to 2045.51] | 1822.43 [1509.74 to 2199.89] | 62.40 [51.85 to 75.08]
  3: number analyzed (Participants) | 164 | 178 | 170 | 178
  3 | 319.33 [263.23 to 387.40] | 407.13 [336.51 to 492.56] | 497.72 [410.26 to 603.84] | 343.29 [283.99 to 414.96]
  4: number analyzed (Participants) | 163 | 176 | 169 | 176
  4 | 1229.24 [1070.97 to 1576.17] | 1717.83 [1419.20 to 2079.30] | 1326.49 [1093.40 to 1609.25] | 1414.77 [1169.79 to 1711.05]
  5: number analyzed (Participants) | 164 | 177 | 170 | 178
  5 | 491.01 [370.31 to 651.05] | 546.38 [413.37 to 722.19] | 366.50 [276.39 to 485.99] | 691.28 [524.10 to 911.78]
  6A: number analyzed (Participants) | 162 | 178 | 170 | 178
  6A | 3252.03 [2439.24 to 4335.64] | 3604.41 [2718.05 to 4779.81] | 3218.37 [2416.99 to 4285.44] | 3932.31 [2969.22 to 5207.78]
  6B: number analyzed (Participants) | 163 | 177 | 170 | 178
  6B | 3506.32 [2730.26 to 4502.96] | 4646.32 [3630.07 to 5947.07] | 4867.77 [3792.29 to 6248.24] | 3783.96 [2961.89 to 4834.20]
  7F: number analyzed (Participants) | 163 | 177 | 165 | 174
  7F | 3318.45 [2768.67 to 3977.40] | 4359.57 [3646.63 to 5211.90] | 5962.25 [4965.38 to 7159.25] | 3975.12 [3324.16 to 4753.56]
  8: number analyzed (Participants) | 164 | 178 | 170 | 178
  8 | 2344.26 [1954.41 to 2811.88] | 2483.57 [2075.88 to 2971.34] | 2668.87 [2224.94 to 3201.37] | 2267.98 [1897.25 to 2711.15]
  9N: number analyzed (Participants) | 162 | 176 | 167 | 172
  9N | 8217.87 [6958.94 to 9704.54] | 9753.78 [8278.27 to 11492.29] | 9066.94 [7672.89 to 10714.27] | 1636.07 [1387.32 to 1929.41]
  9V: number analyzed (Participants) | 164 | 178 | 170 | 177
  9V | 2596.46 [2006.38 to 3360.09] | 3028.18 [2348.52 to 3904.52] | 3757.52 [2903.40 to 4862.91] | 1733.44 [1345.08 to 2233.92]
  10A: number analyzed (Participants) | 161 | 177 | 170 | 176
  10A | 4156.84 [3371.51 to 5125.10] | 5800.54 [4722.94 to 7124.01] | 5366.49 [4358.65 to 6607.37] | 5533.20 [4507.79 to 6791.86]
  11A: number analyzed (Participants) | 164 | 178 | 170 | 177
  11A | 1117.61 [1044.46 to 1195.89] | 1076.79 [1007.27 to 1151.11] | 1064.03 [994.37 to 1138.58] | 1038.01 [971.15 to 1109.47]
  12F: number analyzed (Participants) | 164 | 178 | 170 | 177
  12F | 1550.61 [1187.61 to 2024.56] | 2307.24 [1773.76 to 3001.15] | 1549.29 [1186.52 to 2022.97] | 1914.42 [1472.75 to 2488.55]
  14: number analyzed (Participants) | 163 | 176 | 169 | 177
  14 | 3398.89 [2686.58 to 4300.06] | 4282.68 [3393.98 to 5404.08] | 4107.89 [3246.39 to 5198.01] | 3634.47 [2885.63 to 4577.65]
  15B: number analyzed (Participants) | 163 | 177 | 169 | 177
  15B | 2384.28 [1857.24 to 3060.89] | 3242.54 [2534.98 to 4147.58] | 2535.37 [1975.01 to 3254.71] | 3137.65 [2456.10 to 4008.34]
  17F: number analyzed (Participants) | 164 | 178 | 170 | 171
  17F | 2317.55 [2037.96 to 2635.49] | 2301.19 [2027.23 to 2612.17] | 2290.15 [2013.79 to 2604.43] | 666.74 [586.52 to 757.92]
  18C: number analyzed (Participants) | 163 | 178 | 170 | 177
  18C | 2735.58 [2198.02 to 3404.60] | 3435.80 [2770.54 to 4260.79] | 4103.02 [3298.26 to 5104.14] | 1963.65 [1584.40 to 2433.69]
  19A: number analyzed (Participants) | 164 | 177 | 170 | 178
  19A | 4351.67 [3577.95 to 5292.72] | 5653.21 [4658.23 to 6860.70] | 6211.37 [5106.76 to 7554.90] | 4813.63 [3972.27 to 5833.20]
  19F: number analyzed (Participants) | 164 | 178 | 170 | 178
  19F | 1928.24 [1669.54 to 2227.03] | 2347.67 [2036.83 to 2705.93] | 2453.82 [2124.54 to 2834.14] | 1419.27 [1232.17 to 1634.79]
  20B: number analyzed (Participants) | 164 | 177 | 167 | 168
  20B | 8205.88 [6476.81 to 10396.54] | 8545.04 [6763.81 to 10795.35] | 7809.21 [6150.35 to 9915.50] | 140.23 [110.55 to 177.88]
  22F: number analyzed (Participants) | 163 | 176 | 169 | 176
  22F | 6243.38 [4988.03 to 7814.68] | 7164.92 [5738.17 to 8946.42] | 4843.18 [3869.91 to 6061.23] | 7631.74 [6120.11 to 9516.73]
  23F: number analyzed (Participants) | 164 | 177 | 170 | 177
  23F | 1000.62 [740.33 to 1352.43] | 1368.00 [1015.55 to 1842.76] | 857.41 [634.33 to 1158.95] | 962.52 [715.73 to 1294.42]
  33F: number analyzed (Participants) | 163 | 175 | 169 | 176
  33F | 11672.18 [9582.40 to 14217.70] | 17099.25 [14061.56 to 20793.17] | 11856.15 [9732.71 to 14442.87] | 11030.39 [9085.39 to 13391.78]

7. Secondary Outcome: VAX-24 Pneumococcal Serotype-specific Immunoglobulin G (IgG) Geometric Mean Concentration (GMCs)
Description: Antibody geometric mean concentrations as measured by IgG for the 24 pneumococcal serotypes in VAX-24
Time Frame: 1 month after vaccination
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | VAX-24 Low Dose | VAX-24 Mid Dose | VAX-24 Mixed Dose | PCV20
Number analyzed (Participants) | 166 | 181 | 172 | 179
mcg/mL
  1: number analyzed (Participants) | 164 | 178 | 170 | 178
  1 | 2.85 [2.29 to 3.55] | 4.65 [3.75 to 5.77] | 4.01 [3.22 to 4.99] | 4.39 [3.54 to 5.45]
  2: number analyzed (Participants) | 164 | 178 | 170 | 178
  2 | 13.31 [10.99 to 16.11] | 16.37 [13.56 to 19.76] | 18.73 [15.47 to 22.68] | 1.02 [0.85 to 1.23]
  3: number analyzed (Participants) | 164 | 178 | 170 | 178
  3 | 0.41 [0.34 to 0.50] | 0.53 [0.44 to 0.64] | 0.79 [0.65 to 0.97] | 0.48 [0.40 to 0.59]
  4: number analyzed (Participants) | 164 | 178 | 170 | 178
  4 | 1.79 [1.45 to 2.21] | 2.52 [2.04 to 3.10] | 1.83 [1.48 to 2.26] | 2.02 [1.64 to 2.48]
  5: number analyzed (Participants) | 164 | 178 | 170 | 178
  5 | 2.13 [1.66 to 2.73] | 2.42 [1.90 to 3.10] | 1.78 [1.39 to 2.28] | 3.70 [2.90 to 4.73]
  6A: number analyzed (Participants) | 163 | 178 | 170 | 178
  6A | 3.92 [3.00 to 5.11] | 4.66 [3.59 to 6.06] | 4.38 [3.36 to 5.71] | 4.62 [3.56 to 5.99]
  6B: number analyzed (Participants) | 163 | 178 | 170 | 178
  6B | 2.83 [2.14 to 3.73] | 3.78 [2.87 to 4.97] | 4.43 [3.36 to 5.86] | 2.44 [1.85 to 3.20]
  7F: number analyzed (Participants) | 163 | 177 | 169 | 178
  7F | 4.97 [4.10 to 6.04] | 6.29 [5.20 to 7.61] | 8.82 [7.26 to 10.70] | 4.74 [3.92 to 5.73]
  8: number analyzed (Participants) | 164 | 178 | 170 | 178
  8 | 8.94 [7.25 to 11.02] | 8.79 [7.15 to 10.81] | 8.94 [7.25 to 11.02] | 7.30 [5.95 to 8.97]
  9N: number analyzed (Participants) | 163 | 177 | 169 | 175
  9N | 7.98 [6.72 to 9.48] | 10.78 [9.10 to 12.78] | 7.91 [6.66 to 9.40] | 2.52 [2.13 to 2.99]
  9V: number analyzed (Participants) | 164 | 177 | 169 | 177
  9V | 3.93 [3.13 to 4.92] | 5.12 [4.10 to 6.40] | 7.15 [5.71 to 8.97] | 2.94 [2.36 to 3.67]
  10A: number analyzed (Participants) | 164 | 178 | 170 | 177
  10A | 6.73 [5.30 to 8.54] | 7.90 [6.24 to 10.00] | 6.58 [5.18 to 8.36] | 9.38 [7.41 to 11.86]
  11A: number analyzed (Participants) | 164 | 178 | 170 | 178
  11A | 5.62 [4.73 to 6.67] | 5.76 [4.86 to 6.83] | 4.87 [4.10 to 5.78] | 3.72 [3.14 to 4.40]
  12F: number analyzed (Participants) | 164 | 178 | 170 | 178
  12F | 1.73 [1.40 to 2.15] | 2.13 [1.72 to 2.64] | 1.91 [1.54 to 2.38] | 1.15 [0.93 to 1.42]
  14: number analyzed (Participants) | 164 | 178 | 169 | 178
  14 | 8.62 [6.54 to 11.36] | 10.47 [7.97 to 13.75] | 10.47 [7.93 to 13.81] | 8.17 [6.23 to 10.72]
  15B: number analyzed (Participants) | 163 | 178 | 170 | 178
  15B | 10.67 [8.61 to 13.23] | 14.09 [11.41 to 17.40] | 11.59 [9.36 to 14.36] | 14.81 [12.00 to 18.27]
  17F: number analyzed (Participants) | 164 | 178 | 170 | 178
  17F | 9.57 [7.92 to 11.56] | 10.51 [8.72 to 12.67] | 9.89 [8.18 to 11.95] | 0.46 [0.38 to 0.55]
  18C: number analyzed (Participants) | 164 | 178 | 170 | 178
  18C | 6.66 [5.10 to 8.70] | 8.50 [6.53 to 11.07] | 10.35 [7.92 to 13.53] | 6.67 [5.13 to 8.67]
  19A: number analyzed (Participants) | 163 | 176 | 168 | 176
  19A | 7.35 [5.80 to 9.31] | 9.21 [7.29 to 11.64] | 11.50 [9.07 to 14.58] | 8.84 [7.01 to 11.16]
  19F: number analyzed (Participants) | 164 | 178 | 170 | 178
  19F | 4.98 [3.80 to 6.52] | 8.92 [6.83 to 11.64] | 9.96 [7.60 to 13.04] | 4.34 [3.33 to 5.66]
  20B: number analyzed (Participants) | 163 | 178 | 170 | 177
  20B | 19.53 [16.82 to 22.68] | 24.90 [21.49 to 28.84] | 19.40 [16.71 to 22.52] | 4.06 [3.50 to 4.70]
  22F: number analyzed (Participants) | 164 | 178 | 170 | 178
  22F | 4.13 [3.41 to 5.00] | 5.45 [4.51 to 6.59] | 3.81 [3.15 to 4.61] | 7.32 [6.06 to 8.83]
  23F: number analyzed (Participants) | 164 | 178 | 170 | 178
  23F | 4.60 [3.59 to 5.87] | 5.90 [4.63 to 7.52] | 5.27 [4.12 to 6.73] | 5.18 [4.07 to 6.59]
  33F: number analyzed (Participants) | 163 | 176 | 165 | 175
  33F | 12.20 [10.11 to 14.72] | 17.58 [14.60 to 21.17] | 11.82 [9.77 to 14.30] | 9.73 [8.08 to 11.71]

ADVERSE EVENTS:
Time Frame: 6 months
Description: All subjects had safety labs analyzed at Baseline and Day 29. Solicited AEs were collected for 7 days and unsolicited AEs for 28 days post-vaccination. SAEs, new onset of chronic illness and medically attended adverse events were collected for 6 months post-vaccination. Subject safety data were analyzed according to the vaccine regimen received: 1 subject was randomized to VAX-24 2.2/4.4 mcg but received VAX-24 2.2 mcg, and 2 subjects were randomized to VAX-24 2.2 mcg but received PCV20.
Groups:
- VAX-24 Low Dose 18-49 Yrs; VAX-24 Mid Dose 18-49 Yrs; VAX-24 Mixed Dose 18-49 Yrs; VAX-24 Low Dose 50-64 Yrs; VAX-24 Mid Dose 50-64 Yrs; VAX-24 Mixed Dose 50-64 Yrs; VAX-24 Low Dose 18-64 Yrs; VAX-24 Mid Dose 18-64 Yrs; VAX-24 Mixed Dose 18-64 Yrs: Participants will receive a single dose of VAX-24 administered as an intramuscular injection on Day 1 at one of three dose levels.
  24 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-24 will be administered into the deltoid muscle at Day 1
Arm/Group | VAX-24 Low Dose 18-49 Yrs | VAX-24 Mid Dose 18-49 Yrs | VAX-24 Mixed Dose 18-49 Yrs | PCV20 18-49 Yrs | VAX-24 Low Dose 50-64 Yrs | VAX-24 Mid Dose 50-64 Yrs | VAX-24 Mixed Dose 50-64 Yrs | PCV20 50-64 Yrs | VAX-24 Low Dose 18-64 Yrs | VAX-24 Mid Dose 18-64 Yrs | VAX-24 Mixed Dose 18-64 Yrs | PCV20 18-64 Yrs
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/193 | 0/191 | 0/191 | 0/196 | 0/209 | 0/207 | 0/207 | 0/212
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 2/193 | 3/191 | 1/191 | 4/196 | 2/209 | 3/207 | 1/207 | 4/212
Other Adverse Events (participants affected / at risk) | 9/16 | 13/16 | 14/16 | 16/16 | 161/193 | 155/191 | 164/191 | 163/196 | 170/209 | 168/207 | 178/207 | 179/212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VAX-24 Low Dose 18-49 Yrs (N=16) | VAX-24 Mid Dose 18-49 Yrs (N=16) | VAX-24 Mixed Dose 18-49 Yrs (N=16) | PCV20 18-49 Yrs (N=16) | VAX-24 Low Dose 50-64 Yrs (N=193) | VAX-24 Mid Dose 50-64 Yrs (N=191) | VAX-24 Mixed Dose 50-64 Yrs (N=191) | PCV20 50-64 Yrs (N=196) | VAX-24 Low Dose 18-64 Yrs (N=209) | VAX-24 Mid Dose 18-64 Yrs (N=207) | VAX-24 Mixed Dose 18-64 Yrs (N=207) | PCV20 18-64 Yrs (N=212)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Bladder Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Forearm Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VAX-24 Low Dose 18-49 Yrs (N=16) | VAX-24 Mid Dose 18-49 Yrs (N=16) | VAX-24 Mixed Dose 18-49 Yrs (N=16) | PCV20 18-49 Yrs (N=16) | VAX-24 Low Dose 50-64 Yrs (N=193) | VAX-24 Mid Dose 50-64 Yrs (N=191) | VAX-24 Mixed Dose 50-64 Yrs (N=191) | PCV20 50-64 Yrs (N=196) | VAX-24 Low Dose 18-64 Yrs (N=209) | VAX-24 Mid Dose 18-64 Yrs (N=207) | VAX-24 Mixed Dose 18-64 Yrs (N=207) | PCV20 18-64 Yrs (N=212)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site bruising (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site pain (Skin and subcutaneous tissue disorders) | 9 | 12 | 13 | 13 | 137 | 136 | 147 | 137 | 146 | 148 | 160 | 150
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 3 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 5 | 2 | 1 | 0 | 5
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 4 | 13 | 15 | 17 | 17 | 14 | 16 | 20 | 21
Edema (Skin and subcutaneous tissue disorders) | 3 | 2 | 4 | 3 | 17 | 15 | 15 | 21 | 20 | 17 | 19 | 24
Fatigue (General disorders) | 6 | 5 | 6 | 8 | 82 | 78 | 78 | 78 | 88 | 83 | 84 | 86
Headache (General disorders) | 5 | 6 | 4 | 6 | 59 | 55 | 58 | 59 | 64 | 61 | 62 | 65
Muscle pain (Musculoskeletal and connective tissue disorders) | 6 | 6 | 3 | 9 | 110 | 107 | 115 | 104 | 116 | 113 | 118 | 113
Joint pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2 | 7 | 48 | 31 | 53 | 47 | 52 | 33 | 55 | 54
Fever (General disorders) | 1 | 1 | 0 | 2 | 2 | 1 | 4 | 2 | 3 | 2 | 4 | 4

LIMITATIONS AND CAVEATS:
Some limitations of this clinical study include the lack of a group, such as 3·3 µg or 4·4 µg, for all serotypes, aimed at understanding whether the dose response of polysaccharide can overcome carrier suppression. The relatively low ethnic diversity of participants is also a limitation, which will be addressed in larger phase 3 clinical trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor shall review within the ninety (90) day period. Upon receiving any notification from Sponsor requesting deletion of Confidential Information, correction of inaccuracies, or a delay in publication to allow the filing of patent application, Institution or Investigator shall take the requested action of Sponsor.

DOCUMENTS (2):
  • Study Protocol (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/56/NCT05266456/Prot_002.pdf
  • Statistical Analysis Plan (2022-12-29): https://cdn.clinicaltrials.gov/large-docs/56/NCT05266456/SAP_003.pdf